CLINICAL TRIAL: NCT05248607
Title: Evaluation of the Lived Experience of Overweight/Obese Patients Who Have Benefited From a Mindful Eating Program at Montpellier University Hospital by Semi-structured Face-to-face Interviews.
Brief Title: Lived Experience of Overweight/Obese Patients Who Have Benefited From a Mindful Eating Program.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL22_0073
Record Dates: First submitted 2022-02-07; First posted 2022-02-21 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Overweight or Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to understand the lived experience of overweight/obese patients who have followed the mindful eating program at Montpellier University Hospital. Semi-structured face-to-face interviews will be conducted in the Nutrition-Diabetes service by using a questionnaire.

ELIGIBILITY:
Inclusion criteria:

- People who have attended at least 6 out of 8 sessions of the mindful program

Exclusion criteria:

* People who have attended less than 6 sessions of the program.
* Declining participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited among people who have consulted a doctor in the Nutrition-Diabetes service for overweight/obesity (BMI 25-39.9 kg/m²) and who have followed a mindful eating program led by Béatrix Toto within the service. Each program has 12 participants (2 sessions per year).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Number of participants with the lived experience | day 1
  the experience of overweight/obese patients who have followed the current mindful eating program at Montpellier University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Marion Van Beekum, resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC